CLINICAL TRIAL: NCT04557735
Title: A Phase 3, Open-label, Single Arm, Multicenter Study of Ravulizumab in Addition to Best Supportive Care in Pediatric Participants With Thrombotic Microangiopathy (TMA) After Hematopoietic Stem Cell Transplantation (HSCT)
Brief Title: Study of Ravulizumab in Pediatric Participants With HSCT-TMA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALXN1210-TMA-314; 2020-000761-16 (EudraCT Number)
Record Dates: First submitted 2020-09-02; First posted 2020-09-22 (Actual); Results first posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Thrombotic Microangiopathy
Keywords: Thrombotic Microangiopathy (TMA); Ultomiris; Ravulizumab; Hematopoietic Stem Cell Transplant
MeSH Terms: conditions — Thrombotic Microangiopathies | interventions — ravulizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ravulizumab plus Best Supportive Care (Experimental): Participants will receive ravulizumab plus Best Supportive Care as background therapy.
  Interventions: Drug: Ravulizumab; Other: Best Supportive Care

INTERVENTIONS:
Drug: Ravulizumab — Weight-based doses of ravulizumab will be administered intravenously as a loading dose regimen followed by maintenance dosing every 4 or 8 weeks, depending upon weight.
  Other Names: Ultomiris
Other: Best Supportive Care — Participants will receive medications, therapies, and interventions per standard hospital treatment protocols (unless specifically prohibited by the protocol).

SUMMARY:
This study will evaluate the safety, efficacy, pharmacokinetics, and pharmacodynamics of ravulizumab administered by intravenous infusion to pediatric participants, from 1 month to < 18 years of age, with HSCT-TMA. The treatment period is 26 weeks, followed by a 26-week off-treatment follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 28 days of age up to < 18 years of age at the time of signing the informed consent.
2. Received HSCT within the past 12 months.
3. Diagnosis of TMA that persists for at least 72 hours after initial management of any triggering agent/condition.
4. A TMA diagnosis based on meeting the laboratory-based criteria during the Screening Period and/or ≤14 days prior to the Screening Period.
5. Body weight ≥ 5 kilograms at Screening or ≤7 days prior to the start of the Screening Period (date of consent).
6. Female participants of childbearing potential and male participants with female partners of childbearing potential must use highly effective contraception.
7. Participants must be vaccinated against meningococcal infections if clinically feasible. Participants who cannot receive meningococcal vaccine should receive antibiotic prophylaxis. Participants <18 years of age must be re-vaccinated against Haemophilus influenzae type b (Hib) and Streptococcus pneumoniae if clinically feasible.
8. Participants or their legally authorized representative must be capable of giving signed informed consent or assent.

Exclusion Criteria:

1. Thrombotic thrombocytopenic purpura (TTP) evidenced by ADAMTS13 deficiency.
2. Known Shiga toxin-related hemolytic uremic syndrome as demonstrated by positive test.
3. Positive direct Coombs test indicative of a clinically significant immune-mediated hemolysis not due to TMA.
4. Clinical diagnosis of disseminated intravascular coagulation (DIC).
5. Known bone marrow/graft failure for the current HSCT.
6. Diagnosis of veno-occlusive disease (VOD) which is unresolved at the time of Screening.
7. Human immunodeficiency virus (HIV) infection.
8. Unresolved meningococcal disease.
9. Presence of sepsis requiring vasopressor support.
10. Pregnancy or breastfeeding.
11. Hypersensitivity to murine proteins or to 1 of the excipients of Ravulizumab.
12. Any ongoing or history of medical or psychological conditions unrelated to HSCT-TMA that could increase the risk to the participant or confound the outcome of the study.
13. Respiratory failure requiring mechanical ventilation.
14. Previously or currently treated with a complement inhibitor.
15. Participation in an interventional treatment study of any therapy for TMA.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2024-11-26 (Actual); Study Completion 2025-05-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (8):
  - Research Site, Tucson, Arizona
  - Research Site, Aurora, Colorado
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Portland, Oregon
  - Research Site, Dallas, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Madison, Wisconsin
- Israel (4):
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Petah Tikva
  - Research Site, Ramat Gan
- Research Site, Roma, Italy
- Japan (4):
  - Research Site, Fukushima
  - Research Site, Kobe
  - Research Site, Nagoya
  - Research Site, Osaka
- Research Site, Seoul, South Korea
- Spain (4):
  - Research Site, Barcelona
  - Research Site, Esplugues de Llobregat
  - Research Site, Madrid
  - Research Site, Salamanca
- United Kingdom (3):
  - Research Site, Birmingham
  - Research Site, Bristol
  - Research Site, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ALXN1210-TMA-314&attachmentIdentifier=977d033a-45c7-4d89-bf79-122ac01c1262&fileName=ALXN1210-TMA-314_Final_CSR_Synopsis_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Ravulizumab: Participants received weight-based dosages of ravulizumab intravenously for 26 weeks during the Treatment Period. Participants received a loading dose of ravulizumab intravenously on Days 1, 5 and 10 followed by maintenance dosing on Day 15 and once every 8 weeks or every 4 weeks thereafter depending upon their body weight. After the completion of the treatment period, participants were followed for 26 weeks in Follow-up period (no study drug was administered during this period).
Period: Treatment Period (26 Weeks)
Arm/Group | Ravulizumab
Started | 41
Received at Least 1 Dose of Study Drug | 41
Completed | 29
Not Completed | 12
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 4
Not completed — Death | 5
Not completed — Adverse Event | 2
Period: Follow-Up Period (26 Weeks)
Arm/Group | Ravulizumab
Started | 29
Completed | 24
Not Completed | 5
Not completed — Physician Decision | 1
Not completed — Death | 4

BASELINE CHARACTERISTICS:
Population: Safety set included all participants who signed the informed consent and received at least 1 dose of ravulizumab.
Arm/Group | Ravulizumab
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.6 (5.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 11
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 22
  More than one race | 6
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Participants With Thrombotic Microangiopathy (TMA) Response
Description: The criteria for TMA response were: 1. Normalization of platelet count (defined as platelet count ≥ 50000 mm^3 or >=50% increase in platelet count) without transfusion support during the prior 7 days. 2. Normalization of lactate dehydrogenase (LDH, defined as LDH ≤ upper limit of normal [ULN]) and absence of schistocytes. 3. At least 50% reduction in protein/creatinine ratio from baseline. Participants must meet each TMA criterion at 2 separate assessments obtained at least 24 hours apart, with no criteria failures or more than 1 missed scheduled visit in between. Additionally, all intervals in which the criteria were met must overlap for at least 1 day.
Time Frame: Up to Week 26
Population: Full analysis set included all participants who signed the informed consent and received at least 1 dose of ravulizumab, excluding participants who enrolled prior to availability of shiga toxin-related hemolytic uremic syndrome (ST-HUS) and a disintegrin and metalloproteinase with a thrombospondin type 1 motif, member 13 (ADAMTS13) laboratory results and are subsequently found to be ineligible after enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Ravulizumab
Number analyzed (Participants) | 41
Participants | 7

2. Secondary Outcome: Time to TMA Response During the 26-Week Treatment Period
Description: Time to TMA response was defined as the time from first infusion to the first time point at which all criteria for TMA response was met. Participants were assigned as responders at the time of their TMA response and were censored at the earlier of last assessment with all 3 TMA response components available (including measurements collected after treatment discontinuation), or death if they did not respond by then. TMA response required the following: 1. Normalization of platelet count (defined as platelet count ≥ 50000 mm^3 or >=50% increase in platelet count) without transfusion support during the prior 7 days. 2. Normalization of LDH (defined as LDH ≤ULN) and absence of schistocytes. 3. At least 50% reduction in protein/creatinine ratio from baseline.
Time Frame: Day 1 through Week 26
Population: Full analysis set included all participants who signed the informed consent and received at least 1 dose of ravulizumab, excluding participants who enrolled prior to availability of ST-HUS and ADAMTS13 laboratory results and are subsequently found to be ineligible after enrollment.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Ravulizumab
Number analyzed (Participants) | 41
days | NA [154.0 to NA] — The median and the upper limit of confidence interval could not be reached because fewer than half of the participants experienced an event.

3. Secondary Outcome: Participants With Hematologic Response
Description: Hematologic response required the following: (1) Normalization of platelet count (defined as platelet count ≥ 50000 mm^3 or >=50% increase in platelet count) without transfusion support during the prior 7 days and (2) Normalization of LDH (defined as LDH ≤ULN) and absence of schistocytes.
Time Frame: Up to Week 26
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Ravulizumab
Number analyzed (Participants) | 41
Participants | 10

4. Secondary Outcome: Time to Hematologic Response During the 26-Week Treatment Period
Description: Time to Hematologic response was defined as the time from first infusion to the first time point at which all criteria for hematologic response was met. Participants were assigned as responders at the time of their response and were censored at their discontinuation time or at the end of available follow-up if they did not respond by then. Hematologic response required the following: (1) Normalization of platelet count (defined as platelet count ≥ 50000 mm^3 or >=50% increase in platelet count) without transfusion support during the prior 7 days and (2) Normalization of LDH (defined as LDH ≤ULN) and absence of schistocytes.
Time Frame: Day 1 through Week 26
Population: Full analysis set included all participants who signed the informed consent and received at least 1 dose of ravulizumab, excluding participants who enrolled prior to availability of ST-HUS and ADAMTS13 laboratory results and are subsequently found to be ineligible after enrollment. Here, overall number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Ravulizumab
Number analyzed (Participants) | 41
days | NA [154.0 to NA] — NA signifies that the median and the upper limit of confidence interval could not be reached because fewer than half of the participants experienced an event.

5. Secondary Outcome: Participants With Hemoglobin Response
Description: Hemoglobin response was defined as the ability to maintain hemoglobin ≥ 10 g/dL without RBC transfusion support. The criterion must have been met at 2 separate assessments obtained at least 24 hours apart, and any measurement in between, and without RBC transfusion support during the prior 7 days.
Time Frame: Up to Week 26
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Ravulizumab
Number analyzed (Participants) | 41
Participants | 17

6. Secondary Outcome: Participants With Platelet Response
Description: Normalization of platelet count was defined as baseline platelet count ≤ 50000 mm^3 or > 50000 mm^3, absolute platelet count > 50000 mm^3 or >=50% increase in platelet count without transfusion support during the prior 7 days.
Time Frame: Up to Week 26
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Ravulizumab
Number analyzed (Participants) | 41
Participants | 24

7. Secondary Outcome: Participants With Partial TMA Response
Description: Partial response was defined as a participant meeting at least 1, but not all, criteria for TMA response. TMA response required the following: 1. Normalization of platelet count (defined as platelet count ≥ 50000 mm^3 or >=50% increase in platelet count) without transfusion support during the prior 7 days. 2. Normalization of LDH, (defined as LDH ≤ULN) and absence of schistocytes. 3. At least 50% reduction in protein/creatinine ratio from baseline.
Time Frame: Up to Week 26
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Ravulizumab
Number analyzed (Participants) | 41
Participants | 22

8. Secondary Outcome: Participants With Loss of TMA Response
Description: Loss of response occurred when a participant who had previously achieved a TMA response failed to meet criteria for one or more components of TMA response at a subsequent visit in treatment period. At least one parameter must fail to meet response criteria at 2 separate assessments obtained at least 24 hours apart, and any measurement in between. TMA response required the following: 1. Normalization of platelet count (defined as platelet count ≥ 50000 mm^3 or >=50% increase in platelet count) without transfusion support during the prior 7 days. 2. Normalization of LDH (defined as LDH ≤ULN) and absence of schistocytes. 3. At least 50% reduction in protein/creatinine ratio from baseline.
Time Frame: Up to Week 26
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Ravulizumab
Number analyzed (Participants) | 7
Participants | 2

9. Secondary Outcome: Duration of TMA Response Through Week 52
Description: This analysis includes data for each participant after TMA response through final follow-up. Participants with TMA response who do not experience these events are censored at their end of study date. TMA response required following: 1. Normalization of platelet count (defined as platelet count ≥ 50000 mm^3 or >=50% increase in platelet count) without transfusion support during the prior 7 days. 2. Normalization of LDH (defined as LDH ≤ULN) and absence of schistocytes. 3. At least 50% reduction in protein/creatinine ratio from baseline. The estimate is calculated based on Kaplan-Meier method.
Time Frame: Day 1 through Week 52
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Ravulizumab
Number analyzed (Participants) | 7
days | NA [22.0 to NA] — NA signifies that the median and the upper limit of confidence interval could not be reached because fewer than half of the participants experienced an event.

10. Secondary Outcome: Participants With TMA Relapse
Description: For participants that meet criteria for TMA response during 26-week Treatment Period, TMA relapse is defined as evidence of worsening hematologic and renal dysfunction due to TMA during post-treatment Follow-up Period that requires treatment intervention, as determined by Investigator. TMA response required the following: 1. Normalization of platelet count (defined as platelet count ≥ 50000 mm^3 or >=50% increase in platelet count) without transfusion support during the prior 7 days. 2. Normalization of LDH (defined as LDH ≤ULN) and absence of schistocytes. 3. At least 50% reduction in protein/creatinine ratio from baseline.
Time Frame: Up to Week 52
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Ravulizumab
Number analyzed (Participants) | 7
Participants | 0

11. Secondary Outcome: Overall Survival
Description: The Kaplan-Meier method was used to measure overall survival estimate. Overall survival was calculated from date of treatment start to date of a documented death event (death due to any cause) or date of censoring. Participants who survived were censored at the earliest of an additional hematopoietic stem cell transplant (HSCT), Week 52, or their last known date alive.
Time Frame: Day 1 through Week 52
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Ravulizumab
Number analyzed (Participants) | 41
proportion of participants | 0.734 [0.560 to 0.847]

12. Secondary Outcome: Non-relapse Mortality During the 52-Week Treatment Period
Description: Cumulative incidence was estimated using a competing risk model. Non-relapse mortality was defined as a participant's death due to any cause during the study, with the exception of death due to underlying disease progression or relapse.
Time Frame: Day 1 through Week 52
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Ravulizumab
Number analyzed (Participants) | 41
proportion of participants | 0.184 [0.079 to 0.322]

ADVERSE EVENTS:
Time Frame: Day 1 up to Week 52
Description: Safety set included all participants who signed the informed consent and received at least 1 dose of ravulizumab.
Groups:
- Treatment Period: Ravulizumab: Participants received weight-based dosages of ravulizumab intravenously for 26 weeks during the Treatment Period. Participants received a loading dose of ravulizumab intravenously on Days 1, 5 and 10 followed by maintenance dosing on Day 15 and once every 8 weeks or every 4 weeks thereafter depending upon their body weight.
- Follow-up Period: Ravulizumab: After the completion of the treatment period, participants were followed for 26 Weeks in Follow-up period (no study drug was administered during this period).
Arm/Group | Treatment Period: Ravulizumab | Follow-up Period: Ravulizumab
All-Cause Mortality (participants affected / at risk) | 6/41 | 4/29
Serious Adverse Events (participants affected / at risk) | 30/41 | 15/29
Other Adverse Events (participants affected / at risk) | 41/41 | 23/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Period: Ravulizumab (N=41) | Follow-up Period: Ravulizumab (N=29)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 2 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0
Phimosis (Congenital, familial and genetic disorders) | 1 | 0
Mydriasis (Eye disorders) | 1 | 0
Uveitis (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Multiple organ dysfunction syndrome (General disorders) | 3 | 0
Pyrexia (General disorders) | 2 | 2
Venoocclusive liver disease (Hepatobiliary disorders) | 1 | 0
Graft versus host disease (Immune system disorders) | 1 | 0
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 1 | 0
COVID-19 (Infections and infestations) | 2 | 0
Gastroenteritis clostridial (Infections and infestations) | 2 | 0
Septic shock (Infections and infestations) | 2 | 0
Acinetobacter sepsis (Infections and infestations) | 1 | 0
Adenovirus infection (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Gastroenteritis Escherichia coli (Infections and infestations) | 1 | 0
Gastroenteritis rotavirus (Infections and infestations) | 1 | 0
Gastroenteritis salmonella (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Klebsiella infection (Infections and infestations) | 1 | 0
Mucormycosis (Infections and infestations) | 1 | 0
Norovirus infection (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 1 | 1
Pseudomonal bacteraemia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Stenotrophomonas infection (Infections and infestations) | 1 | 0
Vaginal abscess (Infections and infestations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Seizure (Nervous system disorders) | 3 | 1
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Neurological symptom (Nervous system disorders) | 1 | 0
Partial seizures (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 1
Renal failure (Renal and urinary disorders) | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Stem cell transplant (Surgical and medical procedures) | 1 | 0
Microangiopathy (Vascular disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1
Haemoperitoneum (Gastrointestinal disorders) | 0 | 1
Device related bacteraemia (Infections and infestations) | 0 | 2
Influenza (Infections and infestations) | 0 | 2
Bacterial sepsis (Infections and infestations) | 0 | 1
Device related sepsis (Infections and infestations) | 0 | 1
Ear infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Gonococcal infection (Infections and infestations) | 0 | 1
Pseudomonas infection (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Streptococcal sepsis (Infections and infestations) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Neuroblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Superficial vein thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Period: Ravulizumab (N=41) | Follow-up Period: Ravulizumab (N=29)
Anaemia (Blood and lymphatic system disorders) | 6 (77) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 5 (13) | 1 (1)
Pericardial effusion (Cardiac disorders) | 6 (9) | 0 (0)
Bradycardia (Cardiac disorders) | 3 (3) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 3 (3)
Hypothyroidism (Endocrine disorders) | 3 (3) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 3 (3) | 0 (0)
Ocular hypertension (Eye disorders) | 3 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 10 (14) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 9 (13) | 3 (4)
Vomiting (Gastrointestinal disorders) | 8 (10) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (13) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (6) | 2 (3)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 (6) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Pyrexia (General disorders) | 10 (20) | 6 (11)
Pain (General disorders) | 4 (5) | 2 (2)
Oedema peripheral (General disorders) | 4 (8) | 0 (0)
Fatigue (General disorders) | 3 (3) | 2 (2)
Graft versus host disease in skin (Immune system disorders) | 3 (4) | 0 (0)
Hypogammaglobulinaemia (Immune system disorders) | 3 (4) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 4 (4) | 1 (2)
Staphylococcal infection (Infections and infestations) | 4 (4) | 0 (0)
COVID-19 (Infections and infestations) | 3 (3) | 2 (2)
Sepsis (Infections and infestations) | 3 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 3 (3)
Rhinovirus infection (Infections and infestations) | 1 (1) | 2 (2)
Candida infection (Infections and infestations) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 8 (12) | 1 (4)
Aspartate aminotransferase increased (Investigations) | 7 (12) | 1 (6)
Weight decreased (Investigations) | 3 (3) | 1 (1)
Blood creatinine increased (Investigations) | 3 (11) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 7 (7) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 5 (5) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Headache (Nervous system disorders) | 11 (22) | 3 (3)
Insomnia (Psychiatric disorders) | 3 (3) | 0 (0)
Dysuria (Renal and urinary disorders) | 3 (3) | 0 (0)
Proteinuria (Renal and urinary disorders) | 3 (8) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 4 (7)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0)
Hypotension (Vascular disorders) | 5 (7) | 3 (4)
Hypertension (Vascular disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-09-02): https://cdn.clinicaltrials.gov/large-docs/35/NCT04557735/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-09): https://cdn.clinicaltrials.gov/large-docs/35/NCT04557735/SAP_001.pdf